CLINICAL TRIAL: NCT03662503
Title: Initial Nutritional Strategy and Stature-level Growth During the Neonatal Period of Children Born Moderately Premature: Cohort EPIPAGE 2
Brief Title: Initial Nutritional Strategy and Stature-level Growth During the Neonatal Period of Children Born Moderately Premature
Acronym: EPIPAGE2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-49
Record Dates: First submitted 2018-09-06; First posted 2018-09-07 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Premature Birth
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- nutrition not aggressive group: Children will be grouped according to their calorie and protein during the first week of life. The tertile 1 will represent the group of children with the lowest nutritional intake (called the "nutrition not aggressive ")
- aggressive nutrition group: Children will be grouped according to their calorie and protein during the first week of life. the tertile 3 will define the group of children presenting the contributions highest nutritional levels (called the "aggressive nutrition" group)

SUMMARY:
The growth and nutrition of premature infants during the neonatal period is a concern of neonatology services; it impacts the child's health in the short and long term. The weight deficit, but especially the weak growth of the cranial perimeter during the Neonatal period is associated with an increased risk of long-term neuro-cognitive impairment.

The optimal nutritional strategy, during the neonatal period, of children born moderately premature is not known.

The optimization of nutrition in premature children is therefore a topical issue in neonatology.

Our project aims to evaluate the impact of an aggressive early nutritional strategy characterized by optimized caloric and protein intakes on the stature-level growth of 2000 children born moderately premature GA from 30 WA (week of amenorrhea) to 32 WA + 6 days and included in the national cohort of follow-up of children of small gestational ages.

Nutritional intake during the first week of life will be analyzed in tertile. Children will be grouped according to their calorie and protein during the first week of life. The tertile 1 will represent the group of children with the lowest nutritional intake (called the "nutrition not aggressive "), the tertile 3 will define the group of children presenting the contributions highest nutritional levels (called the "aggressive nutrition" group).

The primary endpoint will be the z-score change in weight, height and head circumference between birth and age (36 adjusted age WA) between the "nonaggressive nutrition" group and the group. "Aggressive nutrition".

The benefits are for public health to harmonize neonatal care practices within a region and to better understand the impact of nutritional strategies on long-term neuro-cognitive development.

DETAILED DESCRIPTION:
The growth and nutrition of premature infants during the neonatal period is a concern of neonatology services; it impacts the child's health in the short and long term. The weight deficit, but especially the weak growth of the cranial perimeter during the Neonatal period is associated with an increased risk of long-term neuro-cognitive impairment.

The optimal nutritional strategy, during the neonatal period, of children born moderately premature is not known.

The optimization of nutrition in premature children is therefore a topical issue in neonatology.

Our project aims to evaluate the impact of an aggressive early nutritional strategy characterized by optimized caloric and protein intakes on the stature-level growth of 2000 children born moderately premature GA from 30 WA to 32 WA + 6 days and included in the national cohort of follow-up of children of small gestational ages.

Nutritional intake (calorie intake and total protein intake) during the first week of life will be analyzed in tertile.

Children will be grouped according to their calorie and protein during the first week of life. The tertile 1 will represent the group of children with the lowest nutritional intake (called the "nutrition not aggressive "), the tertile 3 will define the group of children presenting the contributions highest nutritional levels (called the "aggressive nutrition" group).

The primary endpoint will be the z-score change in weight, height and head circumference between birth and age (36 adjusted age WA) between the "nonaggressive nutrition" group and the group. "Aggressive nutrition".

The benefits are for public health to harmonize neonatal care practices within a region and to better understand the impact of nutritional strategies on long-term neuro-cognitive development.

ELIGIBILITY:
Inclusion Criteria:

* Children born prematurely between 30 WA (week of amenorrhea) and 32 WA + 6 days
* Included in the cohort EPIPAGE 2 with more than 4500 inclusions. The data Perinatal, neonatal and neuro-cognitive outcome at 2 years are available.
* This will include 2,000 children meeting these criteria.

Exclusion Criteria:

* Children with chromosomal abnormalities or malformations congenital
* Children who died during the neonatal period

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Children born prematurely between 30 WA (week of amenorrhea) and 32 WA + 6 days and included in the cohort EPIPAGE 2
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2018-12 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
weight | 36 weeks
  weight in kilograms will be evaluate between birth and age (36 adjusted age SA)
height | 36 weeks
  height in centimeters will be evaluate between birth and age (36 adjusted age SA)
head circumference | 36 weeks
  head circumference in centimeters will be evaluate between birth and age (36 adjusted age SA)

CONTACTS AND LOCATIONS:
Overall Officials: EMILIE GARRIDO PRADALIE, Study Director — APHM
Locations (1):
- Assistance Publique Des Hopitaux de Marseille, Marseille, PACA, France